CLINICAL TRIAL: NCT00154401
Title: Effect of Liraglutide on Glycaemic Control in Subjects With Type 2 Diabetes.
Brief Title: Effect of Liraglutide on Blood Glucose Control in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1571
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: liraglutide

SUMMARY:
This trial is conducted in Europe. The trial is designed to show the effect of treatment with liraglutide or placebo on blood glucose control after 14 weeks in subjects with type 2 diabetes. Liraglutide or placebo is administered by injection once daily in the evening. The trial is a multi-national trial with treatment concealed to participating subjects, investigators and the sponsor. Treatment allocation is random with equal chance of being assigned to each group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with type 2 diabetes mellitus and treated with either diet or single oral drug therapy
* Diet treated subjects: 7.5% < HbA1c < 10%
* Single oral drug therapy subjects: 7.0% < HbA1c < 9.5%
* Body Mass Index (BMI): max 40 kg/m^2

Exclusion Criteria:

* Subjects treated with thiazolidinediones or insulin
* Subjects with any serious medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2005-01; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 14 weeks treatment

SECONDARY OUTCOMES:
Body weight after 14 weeks.
Glycaemic control parameters (fasting plasma glucose, glucose profiles) after 14 weeks.
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (34):
- Denmark (8):
  - Novo Nordisk Investigational Site, Aalborg
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Copenhagen
  - Novo Nordisk Investigational Site, Hellerup
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, Kolding
  - Novo Nordisk Investigational Site, København S
  - Novo Nordisk Investigational Site, Køge
- France (12):
  - Novo Nordisk Investigational Site, Antibes
  - Novo Nordisk Investigational Site, Dax
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Mougins
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Pessac
  - Novo Nordisk Investigational Site, Rennes
  - Novo Nordisk Investigational Site, Vénissieux
- Netherlands (7):
  - Novo Nordisk Investigational Site, 's-Hertogenbosch
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Apeldoorn
  - Novo Nordisk Investigational Site, Groningen
  - Novo Nordisk Investigational Site, Hengelo
  - Novo Nordisk Investigational Site, Sliedrecht
  - Novo Nordisk Investigational Site, The Hague
- Slovakia (7):
  - Novo Nordisk Investigational Site, Banská Bystrica
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Lučenec
  - Novo Nordisk Investigational Site, Prešov
  - Novo Nordisk Investigational Site, Šahy
  - Novo Nordisk Investigational Site, Žilina

REFERENCES:
- [Result] Vilsboll T, Brock B, Perrild H, Levin K, Lervang HH, Kolendorf K, Krarup T, Schmitz O, Zdravkovic M, Le-Thi T, Madsbad S. Liraglutide, a once-daily human GLP-1 analogue, improves pancreatic B-cell function and arginine-stimulated insulin secretion during hyperglycaemia in patients with Type 2 diabetes mellitus. Diabet Med. 2008 Feb;25(2):152-6. doi: 10.1111/j.1464-5491.2007.02333.x. Epub 2008 Jan 14. PMID 18201212
- [Result] Courreges JP, Vilsboll T, Zdravkovic M, Le-Thi T, Krarup T, Schmitz O, Verhoeven R, Buganova I, Madsbad S. Beneficial effects of once-daily liraglutide, a human glucagon-like peptide-1 analogue, on cardiovascular risk biomarkers in patients with Type 2 diabetes. Diabet Med. 2008 Sep;25(9):1129-31. doi: 10.1111/j.1464-5491.2008.02484.x. No abstract available. PMID 19183322
- [Result] Vilsboll T, Zdravkovic M, Le-Thi T, Krarup T, Schmitz O, Courreges JP, Verhoeven R, Buganova I, Madsbad S. Liraglutide, a long-acting human glucagon-like peptide-1 analog, given as monotherapy significantly improves glycemic control and lowers body weight without risk of hypoglycemia in patients with type 2 diabetes. Diabetes Care. 2007 Jun;30(6):1608-10. doi: 10.2337/dc06-2593. Epub 2007 Mar 19. No abstract available. PMID 17372153
- [Result] Horowitz M, Vilsboll T, Zdravkovic M, Hammer M, Madsbad S. Patient-reported rating of gastrointestinal adverse effects during treatment of type 2 diabetes with the once-daily human GLP-1 analogue, liraglutide. Diabetes Obes Metab. 2008 Jul;10(7):593-6. doi: 10.1111/j.1463-1326.2008.00861.x. Epub 2008 Apr 22. No abstract available. PMID 18435773
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com